CLINICAL TRIAL: NCT06877962
Title: The Effect of Home-based Exercise on Postural Abnormalities of Dialysis Patient
Brief Title: The Effect of Home-based Exercise on Postural Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PA25HD-2-02
Record Dates: First submitted 2025-03-05; First posted 2025-03-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: End-Stage Renal Disease; Hemodialysis Complication
Keywords: Tele-exercise; Dialysis Patients; Postural Abnormalities; Balance and Physical Function; Frailty
MeSH Terms: conditions — Kidney Failure, Chronic; Frailty

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocate to intervention group or control group and will be examined in the same way.
Who Masked: Outcomes Assessor
Masking Description: A research project collaborator who is not informed about grouping of participants will obtain outcome measurements of the functional test and postural abnormalities assessments. Outcome adjudicators, and data analysts will be kept blinded to the allocation. Moreover, all investigators, staff, and participants will be kept masked to outcome measurements and trial results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The participants (n = 15) in the study group will be given an online personalized exercise program at home in hemodialysis (HD). Each session will be 40 to 45 min in duration for 3 days per week over 12 weeks, 36 sessions in total.
  Interventions: Behavioral: Home-based Tele Exercise
- Control group (No Intervention): Patients allocated to the control group (n = 15) will receive their standard nephrological care. Through the 12-week period, all control participants will be instructed to maintain the standard treatment regimen and to maintain their customary dietary and physical activity patterns.

INTERVENTIONS:
Behavioral: Home-based Tele Exercise — The participants in the study group will be given an online personalized exercise program at home in hemodialysis (HD) days. Synchronous tele-exercise will be delivered using the free teleconference application (app) (Google Meets software). The groups of tele-exercises will be private, and the professional will send the link for each training session and will control the access of the participants.
  Arms: Exercise group

SUMMARY:
This study evaluates the effects of synchronous home-based tele-exercise on postural abnormalities (FHP and hyper-kyphosis) in dialysis patients. It aims to assess improvements in balance, physical function, and quality of life while reducing fatigue and fall risk.

DETAILED DESCRIPTION:
End-stage renal disease, as one of the serious problems of public health, can significantly influence Musco skeletal system, physical unction and quality of life in dialysis patients. As a result of the treatment limitations, dialysis patients often suffer from postural abnormalities such as hyper-kyphosis and forward head posture (FHP), directly impacting their balance, daily physical activities and fall risk. Such physical issues, coupled with reduced balance and physical capacity can significantly increase the risk of serious injuries such as fractures of hip and spine.

Kyphosis, an abnormal curvature of the spine, result in noticeable changes not only in the pulmonary function but also in the cardiopulmonary capacity. Furthermore, FHP, the forward displacement of the head in the sagittal plane relative to the shoulders, lead to muscular imbalances including the shortening and tightening of the upper trapezius as well as the weakening of the deep flexor muscles of neck around the cervical spine. In addition to affecting body balance and stability, this condition result in a number of problems such as the neck pain, functional disorders and tension headaches. Main factors contributing to those abnormalities include muscular weakness, reduced bone density and a sedentary life style exacerbated by the specific nature of dialysis treatment. Dialysis patients are also at a higher risk of sarcopenia and osteoporosis subsequently affecting their mobility and risk of falls.

Regular exercises, especially home-based ones, could positively influence postural abnormalities and physical function in dialysis patients. Studies have shown that home-based resistance and aerobic exercises improve bone density, standing balance and physical function. Such programs are considered a suitable option for dialysis patients as a result of their ease of implementation as well as the diminished costs associated with visiting the medical centers.

Despite numerous evidence on the positive effect of exercise on dialysis patients, there is not sufficient research on the effect of home-based exercises on hyper-kyphosis and FHP. Particularly, the effect of such programs on dynamic balance require further investigation. Additionally, only a few studies have comprehensively evaluated the weakness and fatigue indicators in these patients.

To improve the effectiveness of home-based exercises, they should be tailored to the patients' personal requirements. These programs can significantly increase the life quality, aerobic capacity and balance indicators despite the challenge of low retention rate.

The investigators hypothesize that synchronous home-based tele-exercise would have a positive impact on reducing the prevalence of physical abnormalities, including FHP and hyper kyphosis, in dialysis patients. The investigators also expect an improvement in their physical function, balance and quality of life while decreasing fatigue.

In this study, the investigators aim to investigate how home-based exercises affect the prevalence of hyper-kyphosis and FHP in dialysis patients. Additionally using standard methods, the investigators evaluate the impact of these abnormalities on patients' balance and physical function and present preventive solutions to reduce fall risks. As for the secondary goals, the investigators aim to evaluate the final effects on quality of life and fatigue indices of hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and over
2. At least 3 months of stable peritoneal dialysis (PD) history
3. Permission from their doctors
4. Have decision-making capacity to enable them to give informed consent to take part in the study
5. Have access to a smart device (e.g., smartphone, laptop or tablet), and have internet access
6. Engaging in physical activity > 3 times per week at moderate to high intensity
7. Participating in regular exercise programs targeting endurance, strength, or flexibility > 3 times per week

Exclusion Criteria:

1. Unstable cardiac status, including angina, decompensated congestive heart failure, or uncontrolled arrhythmias
2. Active infection or acute medical illness
3. Hemodynamic instability
4. Labile glycemic control
5. Individuals unable to exercise entirely, e.g., lower extremity amputations without feasible alternatives for adapted exercise
6. Having severe musculoskeletal pain at rest or with minimal activity
7. Unable to sit, stand or walk unassisted (walking device such as cane or walker allowed)
8. Having shortness of breath at rest or with activities of daily living (NYHAClass IV)
9. Individuals with exercise participation ≥ 3 times per week that addressed ≥ 2 of the domains
10. Myocardial infarction within the past 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Rate of changes in hyper-kyphosis | Pre-test and 3 Months Later (Post-test)
  Evaluating the effect of home-based exercise on hyper-kyphosis using the Debrunner Kyphometer, a non-radiologic gold standard tool. This device measures the kyphosis angle by positioning its arms on the spinous processes of T2-T3 (upper point) and T11-T12 (lower point), with direct angle readings from the calibrated scale. Measurements are taken in degrees, with hyper-kyphosis defined as ≥53° in women and ≥55° in men.
Rate of changes in forward head posture | Pre-test and 3 Months Later (Post-test)
  Evaluating the effect of home-based exercise on forward head posture craniocervical angle (CVA) analysis using digital photogrammetry. Reflective markers are placed on the C7 spinous process and the tragus of the ear, followed by lateral image capture at a standardized 1.5-meter distance. Image analysis software, such as Kinovea, automatically calculates the CVA angle. A normal posture is defined as CVA ≥53°, while a severe forward head posture is <50°.

SECONDARY OUTCOMES:
Rate of changes of balance and fall risk | Pre-test and 3 Months Later (Post-test)
  Assessing balance improvements and fall risk reduction using Timed Up and Go (TUG) Test duration (unit: seconds, Time required to rise, walk 3 meters, turn, and return; diagnostic threshold ≥12 seconds indicates fall risk).
Rate of changes of physical function | Pre-test and 3 Months Later (Post-test)
  Evaluating physical function improvement using the 6-minute walk test (6MWT), which measures the maximum distance covered in 6 minutes (unit: meters). Reference values: 400-700 meters for older adults and 150-346 meters for heart failure patients.
Rate of changes of daily physical activity level | Pre-test and 3 Months Later (Post-test)
  Assessing the effect of home-based exercise on daily activity levels using the LowPAQ questionnaire which evaluates physical activity across occupational, transportation, household, leisure, and sedentary domains, with scoring in MET-minutes per week for light (3.3 MET), moderate (4.0 MET), and vigorous (8.0 MET) activities. Activity levels are categorized as low (<600 MET-min/week), active (600-3000 MET-min/week), and highly active (>3000 MET-min/week), aligned with WHO guidelines.
Rate of changes of fatigue levels | Pre-test and 3 Months Later (Post-test)
  Measuring fatigue levels before and after the intervention using Fatigue Severity Scale (FSS) (9 items on a Likert scale 1-7 (total range 9-63); Score interpretation: ≥36 indicates clinical fatigue, ≤18 indicates no fatigue. ICC = 0.91)
Rate of changes of quality of life | Pre-test and 3 Months Later (Post-test)
  Evaluating improvements in quality of life using the KDQOL-36 questionnaire, which includes SF-12 (general health, reported as a T-score with a mean of 50) and kidney disease-specific subscales: burden of kidney disease (0-100), symptoms and problems (0-100), and effects of kidney disease (0-100). The Kidney Summary Score (KSS) is calculated as the average of the three kidney-specific subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ali Tabibi, Dr, Principal Investigator — Pardis Specialized Wellness Institute
Locations (1):
- Khorshid Dialysis Center, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results reported in the published article will be shared after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the paper is published. No end date
Access Criteria: Not applicable. It will be accessible for public

REFERENCES:
- [Background] Myers J, Chan K, Chen Y, Lit Y, Patti A, Massaband P, Kiratli BJ, Tamura M, Chertow GM, Rabkin R. Effect of a Home-Based Exercise Program on Indices of Physical Function and Quality of Life in Elderly Maintenance Hemodialysis Patients. Kidney Blood Press Res. 2021;46(2):196-206. doi: 10.1159/000514269. Epub 2021 Mar 26. PMID 33774634
- [Background] Jirasirirak S, Disthabanchong S, Ongphiphadhanakul B, Arj-Ong Vallibhakara S, Nimitphong H. Prevalence and predictors of asymptomatic vertebral fracture in patients with end-stage renal disease. Heliyon. 2022 Mar 23;8(3):e09158. doi: 10.1016/j.heliyon.2022.e09158. eCollection 2022 Mar. PMID 35368525
- [Background] Li WY, Chau PH, Dai Y, Tiwari AF. The Prevalence and Negative Effects of Thoracic Hyperkyphosis on Chinese Community-Dwelling Older Adults in Wuhan, Hubei Province, China. J Nutr Health Aging. 2021;25(1):57-63. doi: 10.1007/s12603-020-1441-1. PMID 33367463
- [Background] Yang S, Boudier-Reveret M, Yi YG, Hong KY, Chang MC. Treatment of Chronic Neck Pain in Patients with Forward Head Posture: A Systematic Narrative Review. Healthcare (Basel). 2023 Sep 22;11(19):2604. doi: 10.3390/healthcare11192604. PMID 37830641
- [Background] de Araujo TB, de Luca Correa H, de Deus LA, Neves RVP, Reis AL, Honorato FS, da S Barbosa JM, Palmeira TRC, Aguiar SS, Sousa CV, Santos CAR, Neto LSS, Amorim CEN, Simoes HG, Prestes J, Rosa TS. The effects of home-based progressive resistance training in chronic kidney disease patients. Exp Gerontol. 2023 Jan;171:112030. doi: 10.1016/j.exger.2022.112030. Epub 2022 Nov 21. PMID 36423855
- [Background] Watanabe K, Kamijo Y, Yanagi M, Ishibashi Y, Harada T, Kohzuki M. Home-based exercise and bone mineral density in peritoneal dialysis patients: a randomized pilot study. BMC Nephrol. 2021 Mar 18;22(1):98. doi: 10.1186/s12882-021-02289-y. PMID 33736592
- [Background] Zhang F, Zhou W, Sun Q, Zhai Y, Zhang Y, Su H, Wang Z. Effects of intradialytic resistance exercises on physical performance, nutrient intake and quality of life among haemodialysis people: A systematic review and meta-analysis. Nurs Open. 2021 Mar;8(2):529-538. doi: 10.1002/nop2.274. Epub 2019 Sep 30. PMID 33570280
- [Background] Greenwood SA, Young HML, Briggs J, Castle EM, Walklin C, Haggis L, Balkin C, Asgari E, Bhandari S, Burton JO, Billany RE, Bishop NC, Bramham K, Campbell J, Chilcot J, Cooper NJ, Deelchand V, Graham-Brown MPM, Hamilton A, Jesky M, Kalra PA, Koufaki P, McCafferty K, Nixon AC, Noble H, Saynor Z, Taal MW, Tollit J, Wheeler DC, Wilkinson TJ, Worboys H, Macdonald JH. Evaluating the effect of a digital health intervention to enhance physical activity in people with chronic kidney disease (Kidney BEAM): a multicentre, randomised controlled trial in the UK. Lancet Digit Health. 2024 Jan;6(1):e23-e32. doi: 10.1016/S2589-7500(23)00204-2. Epub 2023 Nov 14. PMID 37968170
- [Background] Lee MK, Lee CJ, Goo SY, Lee TH, Moon JY, Jung J, Kim MJ, Shin SH, Kim JN, Han SN, Lee JE, Lee JY, Chung IM, Jeon JY. Development and application of a home-based exercise program for patients with cardiovascular disease: a feasibility study. BMC Sports Sci Med Rehabil. 2024 Feb 21;16(1):51. doi: 10.1186/s13102-024-00835-3. PMID 38378630
- [Background] Yoo HN, Chung E, Lee BH. The Effects of Augmented Reality-based Otago Exercise on Balance, Gait, and Falls Efficacy of Elderly Women. J Phys Ther Sci. 2013 Jul;25(7):797-801. doi: 10.1589/jpts.25.797. Epub 2013 Aug 20. PMID 24259856